CLINICAL TRIAL: NCT06284785
Title: The Effects of Bariatric Surgery on Kidney Oxygenation in Obese Adults With Type 2 Diabetes and Hyperfiltration
Acronym: ECSTASY
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Dutch Kidney Foundation (Other); Dutch Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Daniel van Raalte, Prof. Dr. Daniel H. van Raalte, Amsterdam UMC, location VUmc
Other Study IDs: 2023.0121
Record Dates: First submitted 2023-08-03; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Kidney Hypoxia; Diabetes Mellitus, Type 2
Keywords: Obesity; Bariatric surgery
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese patients: Obese patients with T2D and hyperfiltration that will undergo bariatric surgery
  Interventions: Procedure: Bariatric surgery
- Healthy controls: Healthy, lean controls with BMI 20-25

INTERVENTIONS:
Procedure: Bariatric surgery — Patients included in our obese patient group are all scheduled to undergo bariatric surgery
  Groups: Obese patients

SUMMARY:
In this study the investigators will examine the effects of VAT reduction by bariatric surgery on kidney hypoxia and compare kidney oxygenation before- and after surgery in both sexes using BOLD-MRI and measures of kidney hemodynamic function. Furthermore, the investigators will assess whether kidney oxygenation is reduced in obese T2D men and women versus various controls as described below. This will determine whether kidney hypoxia can be appointed as a modifiable pathogenic factor in early DKD and non-surgical interventions targeting kidney hypoxia can be designed to slow DKD progression.

DETAILED DESCRIPTION:
DKD (diabetic kidney disease) is the leading cause of chronic kidney disease (CKD) and leading to significant morbidity and early mortality. Although multiple mechanisms underlying DKD have been proposed, the exact underlying mechanisms remain uncertain resulting in limited treatment options. Accumulating evidence, derived from animal and human studies has indicated that chronic kidney hypoxia is a key underlying determinant of DKD and recent studies in T2D patients have related truncal obesity to glomerular hyperfiltration and unfavorable kidney hemodynamic function that may drive kidney hypoxia. Hyperfiltration is defined as increased whole-kidney GFR or as single-nephron hyperfiltration in people with GFR in the normal range. Hyperfiltration is an early recognized key factor driving kidney disease progression in people with diabetes as it drives subsequent eGFR loss. Increased and dysfunctional (i.e., altered adipose tissue biology) visceral adipose tissue (VAT) present in central obesity is thought to disturb the balance between kidney oxygen- consumption and delivery through secretion of endocrine signals resulting in induction of insulin resistance, mitochondrial dysfunction and impaired substrate metabolism amongst others. In line with this theory, reduction of abdominal obesity following bariatric surgery has demonstrated to improve kidney outcomes in some but not in all individuals. In part this may be sex-specific. Since women have a lower risk for progression of DKD, the role of kidney hypoxia in DKD need to be studied in this regard individualized for sex. In this study, the investigators will address the effects of bariatric surgery on changes in kidney oxygenation using a sex-specific approach in people with hyperfiltration.

ELIGIBILITY:
Group 1: T2DM patients with obesity and hyperfiltration

Inclusion criteria:

* Caucasian; man or women aged ≥18 years and <55 years. Females must be pre-menopausal
* Type 2 diabetes mellitus or pre-diabetes with HbA1c ≥45mmol/mol and <10% (<94mmol/mol)
* BMI ≥35
* eGFR>90 ml/min calculated as by CKD-EPI
* Provision of signed and dated, written informed consent prior to any study specific procedures
* Hypertension should be controlled, i.e., ≤ 155/95 mmHg.
* Scheduled for gastric bypass or gastric sleeve

Exclusion criteria:

* Diagnosis of type 1 diabetes mellitus
* Post-menopausal females (defined as no menses >1 year and follicle stimulating hormone (FSH) >31 U/L)
* Cardiovascular disease event in the last 6 months prior to enrollment as assessed by the investigator, including: myocardial infarction, cardiac surgery or revascularization (CABG/PTCA), unstable angina, heart failure, transient ischemic attack (TIA) or significant cerebrovascular disease, unstable or previously undiagnosed arrhythmia.
* Chronic use of sodium-glucose transporter-2 inhibitors, oral glucocorticoids, non-steroidal anti-inflammatory drugs (NSAIDs), immune suppressants, chemotherapeutics, antipsychotics, tricyclic antidepressants (TCAs), diuretics, or monoamine oxidase inhibitors.
* Current urinary tract infection or active nephritis
* History of allergy/hypersensitivity to any of the test agents
* Contra-indication for MRI
* Any other condition that prevents participation as judged by investigator.

Group 2: Non-diabetic lean controls

Inclusion criteria:

* Caucasian; male of female aged ≥18 years and <40 years. Females must be pre-menopausal
* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Normal glucose tolerance confirmed by HbA1c
* No hypertension
* BMI ≥18,5 and <25 kg/m²

Exclusion criteria:

* Macro-albuminuria (defined as UACR>30 mg/mmol)
* Post-menopausal females (defined as no menses >1 year and follicle stimulating hormone (FSH) >31 U/L)*.
* Cardiovascular disease event in the last 6 months prior to enrollment as assessed by the investigator, including: myocardial infarction, cardiac surgery or revascularization (CABG/PTCA), unstable angina, heart failure, transient ischemic attack (TIA) or significant cerebrovascular disease, unstable or previously undiagnosed arrhythmia.
* Chronic use of renin-angiotensin-system blockers, sodium-glucose transporter-2 inhibitors, GLP-1 receptor agonists, DPP-4 inhibitors, oral glucocorticoids, non-steroidal anti-inflammatory drugs (NSAIDs), immune suppressants, chemotherapeutics, antipsychotics, tricyclic antidepressants (TCAs), diuretics ormonoamine oxidase inhibitors.
* Current urinary tract infection or active nephritis
* History of allergy/hypersensitivity to any of the test agents
* Contra-indication for MRI

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants in our patient group will be selected from the Bariatric outpatient clinic.
  Participants in our control group will be selected from the student campus
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Difference in kidney oxygenation before and after bariatric surgery | 1 year
  BOLD-MRI

SECONDARY OUTCOMES:
Difference in kidney oxygenation between men and women | baseline, 1 year
  BOLD-MRI
Difference in kidney oxygenation between obese, hyperfiltering men and women with T2D versus non-diabetic lean controls | Baseline
  BOLD-MRI

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H van Raalte, MD, Principal Investigator — AmsterdamUMC
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No